CLINICAL TRIAL: NCT02464592
Title: Diagnostic Yield and Safety of Transbronchial Lung Biopsy Using Cryoprobes Versus Conventional Forceps. A Multicenter Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Hospital Universitario La Fe (Other); Germans Trias i Pujol Hospital (Other); Hospital General Universitario Santa Lucía (Other); Hospital Universitari de Bellvitge (Other); Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other); Complejo Hospitalario Universitario de Vigo (Other); University of Salamanca (Other); Hospital Universitario de Valladolid (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IIBSP-CRI-2014-05
Record Dates: First submitted 2015-05-06; First posted 2015-06-08 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Lung Diseases, Interstitial
Keywords: Cryoprobes; Transbronchial lung biopsy; Cryobiopsy
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Biopsy with Cryoprobes (Active Comparator): Transbronchial lung biopsy with a cryoprobe.
  Interventions: Procedure: Transbronchial lung biopsy.
- Biopsy with Conventional Forceps (Active Comparator): Transbronchial lung biopsy with conventional forceps.
  Interventions: Procedure: Transbronchial lung biopsy.

INTERVENTIONS:
Procedure: Transbronchial lung biopsy. — Transbronchial lung biopsy with cryoprobe and with conventional forceps.

SUMMARY:
The purpose of this study is to evaluate the diagnostic yield and safety of transbronchial lung biopsies (TBLB) with cryoprobe versus conventional forceps in patients with diffuse lung disease.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Patients with diffuse lung disease candidate to study with transbronchial lung biopsy (TBLB).
* Inform consent signed.

Exclusion Criteria:

* FEV1 <40% of reference value.
* Respiratory insufficiency (pO2 <60 mmHg or pCO2 >45 mmHg).
* Use of anticoagulant therapy or presence of a coagulation (disorder abnormal platelets counts, international normalized ratio > 1.5).
* Bullous emphysema.
* Pulmonary arterial hypertension.
* Hypersensitivity to anaesthetic and sedative drugs (lidocaine, midazolam, propofol, remifentanyl).
* Psychiatric illness.
* Comorbidities that could increase the risk of the TBLB.
* Pregnancy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield of transbronchial lung biopsy (TBLB) | 24 months
  Comparing those TBLB obtained by cryoprobes versus conventional forceps (number of diagnosis with each technique).

SECONDARY OUTCOMES:
Histological quality of samples as defined the presence of alveolar units in each sample. Composite measure. | 24 months
  The quality of samples are defined by the size, presence of artifacts and presence of alveolar units in each sample.
Safety related to the procedure of the TBLB obtained by cryoprobe compared with conventional forceps assessed by chest radiography. | 24 months
  Chest radiography after TBLB.
Safety related to the procedure of the TBLB obtained by cryoprobe compared with conventional forceps assessed by control of bleeding. | 24 months
  Control of bleeding during procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Pajares, PhD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

REFERENCES:
- [Background] Pajares V, Puzo C, Castillo D, Lerma E, Montero MA, Ramos-Barbon D, Amor-Carro O, Gil de Bernabe A, Franquet T, Plaza V, Hetzel J, Sanchis J, Torrego A. Diagnostic yield of transbronchial cryobiopsy in interstitial lung disease: a randomized trial. Respirology. 2014 Aug;19(6):900-6. doi: 10.1111/resp.12322. Epub 2014 Jun 1. PMID 24890124
- [Derived] Pajares V, Nunez-Delgado M, Bonet G, Perez-Pallares J, Martinez R, Cubero N, Zabala T, Cordovilla R, Flandes J, Disdier C, Torrego A; MULTICRIO Group researchers. Transbronchial biopsy results according to diffuse interstitial lung disease classification. Cryobiopsy versus forceps: MULTICRIO study. PLoS One. 2020 Sep 21;15(9):e0239114. doi: 10.1371/journal.pone.0239114. eCollection 2020. PMID 32956379